CLINICAL TRIAL: NCT07142499
Title: A Pilot of Memory Support System for Older Chinese Americans With Mild Cognitive Impairment
Brief Title: Memory Support System for Older Chinese Americans With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Clara Li, Associate Professor of Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 22-1738
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSS Intervention Group (Experimental): 10-session MSS Training Workbook. Additional sessions beyond the standard 10 sessions can be added up to a maximum of 15 total sessions.
  Interventions: Behavioral: Memory Support System
- Brain Health Education Control Group (Active Comparator): 10 session Brain Health Education. Additional sessions beyond the standard 10 sessions can be added up to a maximum of 15 total sessions.
  Interventions: Behavioral: Brain Health Education

INTERVENTIONS:
Behavioral: Memory Support System — Participants and study partners in the MSS treatment group will work with a study trainer to learn the MSS and eventually adapt the skills to support functioning in their daily life. The MSS trainer will follow a 10-session MSS Training Workbook as the standardized protocol for training. Additional sessions beyond the standard 10 sessions can be added if needed to support mastery of the MSS (up to a maximum of 15 total sessions). Participants and study partners will also receive a copy of the brain health education workbook that contains the same educational information for the control group at the 8-week follow up.
  Other Names: MSS
  Arms: MSS Intervention Group
Behavioral: Brain Health Education — Participants and study partners in the control group will be provided with the MSS guidebook and day planner for self-study of the MSS system. They will also meet with a study trainer to complete 10 sessions of a brain health education course that is tailored for individuals with MCI. The trainer will use a HABIT-based brain health education workbook to provide the content. Additional sessions beyond the standard 10 sessions can be added up to a maximum of 15 total sessions. Participants and study partners will receive a copy of the brain health education workbook at the 8-week follow up.
  Arms: Brain Health Education Control Group

SUMMARY:
The Memory Support System (MSS) from the Healthy Action to Benefit Independence & Thinking® (HABIT) Program is an evidence-based, non-pharmacological intervention for mild cognitive impairment (MCI). Despite the clinical benefits and feasibility, the MSS was primarily developed and used with non-Hispanic White, English-speaking adults. Racial/ethnic minority groups are chronically under-enrolled in clinical trials for Alzheimer's Disease and Alzheimer's Disease Related Dementias (AD/ADRD) due to lack of linguistically and culturally appropriate adaptation of assessment measures and intervention protocols. The purpose of this research study is to examine whether the MSS from HABIT can help Chinese American older adults with mild thinking and memory problems. Target recruitment is 60 Chinese American adults who are primarily Mandarin- (n=30) and Cantonese-speaking (n=30). Forty participants will participate in the trainer-led day planner training and 20 will participate in self-study of the day planner and receive brain health education. Each participant will also be asked to identify a study partner to participate with them.

ELIGIBILITY:
Inclusion criteria:

* self-identify as Chinese American;
* age 55 and above;
* a diagnosis of MCI as confirmed through documented clinical assessment and/or research-based diagnostic criteria;
* predominantly Cantonese- or Mandarin-speaking;
* able to read and write in Chinese;
* visual and auditory acuity adequate for cognitive testing;
* willing to complete the assessment measures;
* having someone in regular contact to serve as a study partner/informant;
* absence or stable use of prescribed memory-enhancing medications within the last 3 months.

Exclusion criteria include:

* any significant neurologic disease that would impact their participation and completion of the trial;
* history of psychiatry disorder (DSM 5 criteria) within the last 12 months;
* history of reading or writing disability sufficient to interfere with MSS training; or
* concurrent participation in another relevant clinical trial.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | baseline, week 1 of intervention session
  Recruitment rate will be measured by dividing the number of enrollees over the number of total potential participants approached.
Retention rate | baseline, treatment end (4-9 weeks)
  Retention rate will be measured by dividing the number of enrollees who remain in the study over the total number of enrollees.
Completion rate | baseline, treatment end (4-9 weeks)
  Completion rate will be measured by dividing the number of enrollees who complete all study procedures over the number of total enrollees.

SECONDARY OUTCOMES:
Everyday Cognition questionnaire | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Functional status will be assessed using selected items from the informant-rated version of the Everyday Cognition (ECog) questionnaire to evaluate a participant's ability to perform everyday tasks in areas of memory and executive functioning.
  Full ECog is comprised of 39 items, each item score 1-4. Total score range from 39-156, with higher score indicating poorer health outcome.
Functional Activities Questionnaire (FAQ) | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  The FAQ, consisting of 10 items assessing instrumental activities of daily living (IADLs), is an informant-based questionnaire, to evaluate functional abilities. The min score is 0 and max score is 30. A higher score generally indicates poorer functioning and ability to perform daily activities.
The Pillbox Test | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  The pillbox Test will also be used to assess performance based IADLs, min score is 0 and max score is 5. A higher score on the pillbox test typically indicates better cognitive function and medication management skills.
Dementia Rating Scale-2 (DRS-2) | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Cognition will be measured using the Dementia Rating Scale-2 (DRS-2). The assessment provides quantitative assessment on attention, initiation/perseveration, construction, conceptualization, and memory. Full score range from 0-144, with higher score indicating better health outcome. It will be used to assess whether treatment group participants demonstrate improved cognitive performance beyond expected practice effect in comparison to their control group counterparts.
Chronic Disease Self-Efficacy Scales | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Self-efficacy for memory will be assessed using modified, selected items from the Chronic Disease Self-Efficacy Scales. Total scores range from 9 to 90, with higher scores indicating greater memory self-efficacy.
Quality of Life in Alzheimer Disease | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Quality of life will be measured using the Quality of Life in Alzheimer Disease instrument, a 13-item measure that has been utilized in MCI and with study partners to assess health-related quality of life. Quality of life of both participant and study partner will be assessed. Total score range 13-52, with higher scores indicating greater quality of health.
Neuropsychiatric Inventory Questionnaire (NPI-Q) - Severity | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Neuropsychiatric symptoms will be assessed using the Neuropsychiatric Inventory Questionnaire (NPI-Q). The instrument is completed by a study partner in which a series of questions are described to assess 12 neuropsychiatric symptoms. If the symptom is present within the last month, the study partner will then rate the severity levels using a 3-point Likert scale (1=mild; 2=moderate; 3= severe).
  Total score range from 12-36, with higher score indicating greater severity.
Center for Epidemiologic Studies Depression Scale | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Depression will be measured using the Center for Epidemiologic Studies Depression Scale, a 20-item self-report scale with 3-point Likert-type response options ranging from 1 (rarely or none of the time or < 1 day) to 3 (most or all of the time or 5-7 days). Total scores range from 0 to 60, with higher scores suggesting greater symptoms of depression. Depression symptomology of both participant and study partner will be assessed.
Anxiety Inventory Form | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Anxiety will be measured using the Anxiety Inventory Form, a 10-item rating scale modified from the State- Trait Anxiety Inventory by the Resources for Enhancing Alzheimer's Caregiver Health project. Total scores range from 10 to 40, with higher scores indicating higher levels of anxiety. Anxiety symptomology of both participant and study partner will be assessed.
Pittsburgh Sleep Quality Index | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Quality and patterns of sleep will be measured with the Pittsburgh Sleep Quality Index, with total scores ranging from 0 to 21; a total score of 5 or greater is indicative of poor sleep. Sleep quality of both participant and study partner will be assessed.
Caregiver Burden Inventory Short-Form | at baseline, treatment end (4-9 weeks), and 8-week follow-up
  Caregiver burden will be assessed by the Caregiver Burden Inventory Short-Form, a 12-question inventory that measures the degree of stress experienced by caregivers concerning the effect of the participant's disability on care partners' lives. Total score range from 0-48, with higher score indicating higher burden

CONTACTS AND LOCATIONS:
Overall Officials: Clara Li, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Li Lab, Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Information will be only shared within the research team at ISMMS, and with collaborators: Dr. Joyce Tam at Rush University Medical Center.